CLINICAL TRIAL: NCT03323944
Title: Phase I Study of Human Chimeric Antigen Receptor Modified T Cells (CAR T Cells) in Patients With Pancreatic Cancer
Brief Title: CAR T Cell Immunotherapy for Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 827644 (UPCC 14217)
Record Dates: First submitted 2017-10-19; First posted 2017-10-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Cancer of the Pancreas
Keywords: metastatic adenocarcinoma, pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: huCART-meso cells via intravenous infusion (IV). (Experimental): Subjects will receive a single dose of 1-3x10^7/m^2 lentiviral transduced huCART-meso cells on day 0 via intravenous infusion.
  Interventions: Biological: huCART-meso cells
- Cohort -1: low dose huCART-meso cells via intravenous infusion (Experimental): In the event that 2 DLTs occur among subjects enrolled in Cohort 1, then enrollment in Cohort 1 will be stopped and the dose will be de-escalated by 10-fold to 1-3x10^6 cells/m^2. Subjects will receive a single dose of 1-3x10^6 cells/m^2 lentiviral transduced huCART-meso cells on day 0.
  Interventions: Biological: huCART-meso cells
- Cohort 2 - huCART meso cells via intraperitoneal infusion (IP) (Experimental): Permanently closed
  Interventions: Biological: huCART-meso cells
- Cohort 3 - huCART meso cells via intrahepatic infusion (hepatic arterial infusion) (Experimental): Permanently closed
  Interventions: Biological: huCART-meso cells
- Cohort 4 - huCART meso cells via intrahepatic infusion (hepatic arterial infusion) (Experimental): Subjects will receive a single dose of of 1-3x10^7 cells/m^2 lentiviral transduced huCART-meso cells on day 0 following a minimum 1 week washout from standard care chemotherapy. This initial intrahepatic infusion may be followed by up to two additional infusions of huCART-meso cells via intravenous (IV) administration at the same dose level, given between 21-42 days apart.
  Interventions: Biological: huCART-meso cells

INTERVENTIONS:
Biological: huCART-meso cells — Intravenous administration or local delivery of lentiviral transduced huCART-meso cells.

SUMMARY:
Phase I study to establish the safety and feasibility of both intravenous administration and local delivery of lentiviral transduced huCART-meso cells in patients with histologically confirmed unresectable or metastatic pancreatic adenocarcinoma

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety and feasibility of lentiviral transduced huCART-meso cells in up to 4 cohorts. Lymphodepleting chemotherapy will not be utilized as part of the planned dosing strategy.

• Cohort 1 (N=3-6): will receive a single dose of 1-3x10^7/m^2 lentiviral transduced huCART-meso cells on day 0 via intravenous infusion.

* Enrollment into Cohort 1 will be paused after the 3rd subject is infused to allow for a formal DLT assessment (performed by the Clinical PI and Medical Director) and DSMB review. If 1 DLT/3 subjects occurs in Cohort 1, the Sponsor (with guidance from the DSMB), will determine whether the study will enroll an additional 3 subjects at this dose level to further establish safety via intravenous infusion, or advance to Cohorts 2 and 3 to explore local delivery of huCART-meso cells at the same dose level. If 0 DLT/3 subjects or 1 DLT/6 subjects occurs at any time, the study may advance to Cohorts 2 and 3.
* If 2 DLTs occur at this dose level at any time, enrollment in Cohort 1 will be stopped and the dose will be de-escalated by 10-fold to 1-3x10^6 cells/m^2 (Cohort -1).
* The infusions in Cohort 1 will be staggered by at least 28 days to allow for the assessment of DLTs for cohort progression, expansion, or dose de-escalation.

In the event that 2 DLTs occur among subjects enrolled in Cohort 1, then enrollment in Cohort 1 will be stopped and the dose will be de-escalated by 10-fold to 1-3x10^6 cells/m^2. This de-escalated cohort will be designated Cohort -1.

• Cohort -1 (N=3-6): will receive a single dose of 1-3x10^6 cells/m^2 lentiviral transduced huCART-meso cells on day 0. Up to 6 subjects will be infused in Cohort -1 if ≤ 1 DLT occurs.

If 0 DLT/3 subjects or 1 DLT/6 subjects occurs in Cohort 1, the study will advance to allow for additional cohorts to be explored.

* Cohorts 2 and 3. Enrollment into these additional cohorts may occur in parallel, however infusions will be staggered as follows to allow for monitoring/assessment of toxicities:
* Cohorts 2 and 3: As of Protocol Amendment V7, Infusion #1/Day 0 for the next 6 subjects in Cohorts 2 and 3 must be staggered by at least 28 days; This includes a minimum of 3 evaluable subjects in Cohort 2 and 3 evaluable subjects in Cohort 3. A DLT assessment will be performed after the 3rd evaluable subject in each cohort reaches the Day 21 safety follow-up visit. If no DLTs are identified in the 1st three evaluable subjects in both Cohorts 2 + 3, subsequent infusions of new subjects within either cohort may occur in parallel; however, no more than two new subjects may be infused within a 14-day period, irrespective of cohort assignment. If both cohorts have not yet infused 3 evaluable subjects without a DLT, all infusions will continue to be staggered by 28 days until this provision is met.
* Cohort 4: Infusion #1/Day 0 for the first 3 subjects in Cohort 4 must be staggered by at least 28 days. A DLT assessment will be performed after the 3rd evaluable subject in this cohort reaches the Day 21 safety follow-up visit. If no DLTs are identified in the 1st three evaluable subjects, subsequent infusions of new subjects may occur in parallel, however no more than two new subjects may be infused within a 14-day period. If 1 DLT is identified in the 1st three evaluable subjects, Infusion #1 for all subsequent subjects will continue to be staggered by at least 28 days and DLT assessments will be performed after each evaluable subject reaches the Day 21 safety follow-up visit.

  * Cohort 2 Participants (N = Up to 6): will receive a single dose of 1-3x10^7/m^2 lentiviral transduced huCART-meso cells on day 0 via intraperitoneal (i.p.) administration. The initial i.p. infusion may be followed by up to two additional infusions of huCART-meso cells via intravenous (IV) administration at the same dose level, given between 21-42 days apart. The subject must meet eligibility to receive additional infusions.

**Cohort 2 is prematurely closed. This closure is the result of feasibility concerns specific to the clinical/disease status of these patients at this stage of their treatment.**

• Cohort 3 Participants (N = Up to 6): will receive a single dose of 1-3x10^7/m^2 lentiviral transduced huCART-meso cells on day 0 via intrahepatic delivery (Hepatic Arterial Infusion). The initial intrahepatic infusion may be followed by up to two additional infusions of huCART-meso cells via intravenous (IV) administration at the same dose level, given between 21-42 days apart. The subject must meet eligibility to receive additional infusions.

**Cohort 3 is prematurely closed. This closure is the result of feasibility concerns specific to the clinical/disease status of these patients at this stage of their treatment.**

• Cohort 4 Participants (N = Up to 6): will allow for the administration of lentiviral transduced huCART-meso cells during 1st line standard of care chemotherapy. A single dose of 1-3x10^7/m^2 huCART-meso cells will be administered on day 0 via intrahepatic delivery (Hepatic Arterial Infusion), following a 1 week washout after standard of care chemotherapy. This initial intrahepatic infusion may be followed by up to two additional infusions of huCART-meso cells via intravenous (IV) administration at the same dose level, given between 21-42 days apart. The subject must meet all eligibility to receive additional infusions. Additional doses of standard of care chemotherapy may also be administered between huCART-meso infusions at the physician-investigator's discretion, as long as the required washout windows are appropriately adhered to. huCART-meso infusions may also be discontinued at any time in favor of resuming standard of care chemotherapy at the physician-investigator's discretion.

Adverse events will be collected and evaluated during the protocol specified adverse event reporting period. Subjects will be continually evaluated for dose-limiting toxicities (DLT). In the event of 2 DLTs in a specific cohort, additional enrollment and treatment activity will be paused to allow for further investigation.

ELIGIBILITY:
* Inclusion Criteria

  1. Patients with the following diagnoses:

     1. Cohorts 1 and -1: Histologically confirmed unresectable or metastatic pancreatic adenocarcinoma
     2. Cohort 2: Histologically confirmed unresectable or metastatic pancreatic adenocarcinoma; and either cytologically-proven ascites or known peritoneal disease on radiologic imaging.
     3. Cohort 3 - 4: Histologically confirmed unresectable or metastatic pancreatic adenocarcinoma with liver metastases as confirmed by pathology or radiographic imaging.
  2. INCLUSION CRITERIA HAS BEEN RETIRED
  3. Prior treatment requirements:

     1. Cohorts 1 - 3: Failure of at least one prior standard of care chemotherapy for advanced stage disease.
     2. Cohort 4: At lease stable disease on the first-line standard of care chemotherapy for advanced stage disease.
  4. Cohorts 1-3 and -1: Subjects must have measurable disease as defined by RECIST 1.1 criteria.
  5. Patients ≥ 18 years of age.
  6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  7. Satisfactory organ and bone marrow function as defined by the following:

     i. Absolute neutrophil count ≥ 1,000/μl ii. Platelets ≥75,000/μl iii. Hemoglobin ≥ 8 g/dL iv. Direct bilirubin ≤ 2.0 mg/dl unless the subject has Gilbert's disease syndrome (≤ 3.0 mg.dl) v. Creatinine ≤ 1.5x the institutional normal upper limit vi. Albumin ≥ 2 vii. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤5x the institutional normal upper limit viii. Cardiac ejection fraction of ≥40% as measured by resting echocardiogram, with no clinically significant pericardial effusion.
  8. Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤ 1.5 and a PTT ≤ 1.2 time the upper limit of normal unless the patient is therapeutically anti-coagulated for history of cancer-related thrombosis and has stable coagulation parameters.
  9. Provides written informed consent.
  10. Subjects of reproductive potential must agree to use acceptable birth control methods
* Exclusion Criteria:

  1. EXCLUSION CRITERIA HAS BEEN RETIRED
  2. Active invasive cancer other than pancreatic adenocarcinoma. Patients with active non-invasive cancers (such as non-melanoma skin cancer, superficial cervical and bladder cancer, or prostate cancer with PSA level < 1.0) are not excluded.
  3. HIV infection
  4. Active hepatitis B or hepatitis C infection
  5. Active autoimmune disease (including but not limited to: systemic lupus erythematosus, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) requiring immunosuppressive therapy within 4 weeks prior to eligibility confirmation by physician-investigator, with the exception of thyroid replacement.
  6. Patients with ongoing or active infection.
  7. Dependence on systemic steroids or immunosuppressant medications.
  8. Patients requiring supplemental oxygen therapy.
  9. Prior therapy with lentiviral gene modified cells.
  10. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
  11. Any clinically significant pericardial effusion, Class II-IV cardiovascular disability according to the New York Heart Association Classification or other cardiovascular condition that would preclude assessment of mesothelin induced pericarditis or that may worsen as a result of toxicities expected for this study. This determination will be made by a cardiologist if cardiac issues are suspected.
  12. Any clinically significant pleural or peritoneal effusion that cannot be drained with standard approaches. An indwelling drainage device placed prior to eligibility confirmation by physician-investigator is acceptable.
  13. Pregnant or breastfeeding women.
  14. EXCLUSION CRITERIA HAS BEEN RETIRED
  15. EXCLUSION CRITERIA HAS BEEN RETIRED
  16. Patients with significant lung disease as follows:

  <!-- -->

  1. Patients with radiographic evidence of greater than lobar lymphangitic pulmonary involvement, greater than lobar bronchial wall thickening suggestive of peribronchial lymphatic disease extension, and/or evidence of extensive bilateral parenchymal metastatic burden. Note: "Greater than lobar" = "in more than 1 lobe".
  2. Patients with radiographic and/or clinical evidence of active radiation pneumonitis.
  3. Patients with radiographic evidence of underlying interstitial lung disease, including evidence of unresolved drug toxicity from any agent (e.g. chemotherapy, targeted agents, amiodarone, nitrofurantoin, etc)
  4. Patients with radiographic evidence of significant pleural effusion that is not readily amenable to minimally invasive drainage.

  17. Cohort 3 and 4 Subjects Only: Patients with a contraindication to IV contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Number of study subjects with treatment-related adverse events using NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.03 | 2 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
Overall survival (OS) | 2 years
Objective response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark O'Hara, MD, Principal Investigator — Assistant Professor of Medicine, Penn Medicine
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Aznar MA, Good CR, Barber-Rotenberg JS, Agarwal S, Wilson W, Watts A, Zhang Z, Gonzales D, Donahue G, Hwang WT, Rennels AK, Rech AJ, Kuramitsu S, Huang H, Glastad KM, Alexander KA, Plesa G, Dowd E, Brennan A, Siegel DL, Tanyi J, Haas A, Torigian DA, Nadolski G, Gonzalez VE, Hexner EO, Fraietta JA, Jadlowsky JK, Young RM, Berger SL, June CH, O'Hara MH. Clinical and molecular dissection of CAR T cell resistance in pancreatic cancer. Cell Rep Med. 2025 Sep 16;6(9):102301. doi: 10.1016/j.xcrm.2025.102301. Epub 2025 Aug 18. PMID 40829595